CLINICAL TRIAL: NCT03307629
Title: NOX66 and Palliative Radiotherapy in Patients With Late-Stage Prostate Cancer - a Phase 1b Proof of Concept and Dose Confirmation Study
Brief Title: Safety and Tolerability of NOX66 in Combination With Palliative Radiotherapy in Patients With Late-Stage Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noxopharm Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOX66-002A
Record Dates: First submitted 2017-09-27; First posted 2017-10-12 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOX66 + Radiation treatment (combined) in cohorts 1-3 (Experimental): NOX66 administered on Days 1-16 and radiation treatment given on Day 2 to 9 of 2-week cycle.
  NOX66 treatment given to 3 cohorts of 4 patients as 1 of 3 doses, 400mg, 800mg and 1200 mg.
  Radiation treatment of 20Gy given over 5 daily fractions to selected target lesion/s for all cohorts.
  Interventions: Drug: NOX66; Radiation: Irradiation Therapy
- NOX66 + Radiation treatment (combined) in cohort 4 (Experimental): NOX66 administered on Days 1-16 and radiation treatment given on Day 2 to 9 of 2-week cycle.
  NOX66 dose will be either one of 3 doses 400mg, 800mg and 1200 mg based on interim analyses of safety data and tumour response at WEEK 6 of 3 dose cohorts of 12 total patients. The Safety Steering Committee will inform on dose for cohort expansion.
  Radiation treatment of 20Gy given over 5 daily fractions to selected target lesion/s for all cohorts.
  Interventions: Drug: NOX66; Radiation: Irradiation Therapy

INTERVENTIONS:
Drug: NOX66 — NOX66 delivered as rectal suppository.
Radiation: Irradiation Therapy — Radiation per selected tumour lesion.

SUMMARY:
The study is intended as a Proof of Concept and dose confirmation study. The primary objective of this study is to observe safety and tolerability of idronoxil (NOX66) in combination with radiotherapy (at palliative doses) in patients with metastatic castrate-resistant prostate cancer (CRPC) and to confirm dose in order to progress to Phase 2/3.

DETAILED DESCRIPTION:
This study will investigate three escalating doses of NOX66 in combination with palliative dose of radiation therapy to establish safety profile and / or obtain efficacy signals and to determine the optimal dose for future radiation therapy combination studies.

The key hypotheses to be tested in this study are:

1. That NOX66 can be safely added to palliative dose radiation therapy.
2. That NOX66 may sensitise tumours to palliative doses of radiation therapy
3. That NOX66 in combination with radiation therapy may trigger or augment an abscopal effect

Participants will have a minimum of 1 symptomatic lesion amenable to radiation therapy.

Radiation therapy will be delivered at a 20Gy dosage over 5 fractions. NOX66 will be taken on 13 consecutive days starting 1 day prior to radiotherapy.

The response of irradiated and non-irradiated target tumour lesions will be measured by CT/MRI scan and RECIST1.1 criteria at three time points post treatment. Pain response will be evaluated using the Brief Pain Inventory-Short Form (BPI-SF) instrument at five time points post treatment.

Patients will be suitable for the study as they become indicated for palliative radiation therapy for management of their cancer.

This study will enrol up to 24 patients in 3 NOX66 dose level cohorts of 4 patients (n=12) and an expansion cohort of 12 patients. Dose escalation decisions will be based on patients who experience adverse events directly related to NOX66 treatment.

Following the review of accumulated safety data, disease status and treatment efficacy signals at WEEK 6 for the first 12 patients, the Study Steering Committee will determine the dose at which to continue treatment for the expansion patient Cohort 4 in the study. A further 12 patients will be recruited at this dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. ≥ 18 years of age
3. Histologically confirmed prostate cancer and/or PSA of >100 ng/mL at original diagnosis
4. Metastatic disease evidenced by either CT/MRI imaging or bone scan
5. Objective evidence of disease progression as defined by either:

   i. Radiographic progression of in nodal or visceral metastases and bone disease progression with 2 or more new lesions ii. Rising PSA value ≥2ng/ml in at least 3 measurements, at least 1 week apart, with castrate levels of serum testosterone.
6. Eligible to receive palliative radiation therapy for management of disease
7. At least one symptomatic lesion which is suitable for radiation therapy
8. ECOG Performance status 0-2
9. A minimum life expectancy of 24 weeks
10. Adequate bone marrow, hepatic and renal function as evidenced by:

    * Absolute neutrophil count (ANC) > 1.5 x 109/L
    * Platelet count > 100 x 109/L
    * Hemoglobin > 9.0 g/dL
    * Serum bilirubin < 1.5 x ULN
    * AST/ALT (SGOT/SGPT) < 2.5 x ULN for the reference laboratory or < 5 x ULN in the presence of liver metastases
    * Serum creatinine < 1.5 x ULN
11. Ongoing androgen deprivation therapy with luteinizing hormone-releasing hormone (LHRH) agonist or antagonist
12. At least 4 weeks must have elapsed prior to commencement of NOX66 treatment since prior chemotherapy, investigational drug or biologic therapy and any toxicity associated with these treatments has recovered to ≤ NCI-CTCAE (version 4.03) Grade 1.
13. At least 21 days must have elapsed following major surgery and any surgical incision should be completely healed.

Exclusion Criteria:

1. Tumour involvement of the central nervous system
2. Uncontrolled infection or systemic disease
3. Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease, angina, and cardiac arrhythmias) or myocardial infarction within the last 12 months

   • Patients with a QTc > 470 msec on screening ECG
4. Concurrent systemic chemotherapy or biological therapy
5. Any situation where the use of suppository therapy is contra-indicated or impractical (eg. chronic diarrhoea, colostomy, ulcerative colitis).
6. Known human immunodeficiency virus (HIV) or Hepatitis B or C (active, previously treated or both)
7. Any subject whose testosterone is not suppressed i.e. is > 0.5nmols/L
8. Any other reason which, in the opinion of the investigator, will preclude suitable participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marinella Messina, PhD, Study Chair — Noxopharm Limited
Locations (10):
- Australia (5):
  - Genesis Cancer Care - Newcastle, Newcastle, New South Wales
  - Central West Cancer Care Centre - Orange Health Service, Orange, New South Wales
  - Genesis Cancer Care Mater Hospital, Sydney, New South Wales
  - North West Cancer Centre, Tamworth Hospital, Tamworth, New South Wales
  - Radiation Oncology Centres Gold Coast, Gold Coast, Queensland
- Georgia (4):
  - Research Institute of Clinical Medicine, Tbilisi
  - TSMU The First University Clinic, Tbilisi
  - National Center of Urology, Tbilisi
  - Institute for Personalised Medicine, Tbilisi
- Canterbury Urology Research Trust, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measure will be made available within 12 months after study completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after study completion

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - NOX66 400mg Daily: NOX66 administered on Days 1-16 and radiation treatment given on Day 2 to 9 of 2-week cycle.
  NOX66 dose of 400mg daily.
  Radiation treatment of 20Gy given over 5 daily fractions to selected target lesion/s for all cohorts.
  NOX66: NOX66 delivered as rectal suppository.
  Irradiation Therapy: Radiation per selected tumour lesion.
- Cohort 2 - NOX66 800mg Daily: NOX66 administered on Days 1-16 and radiation treatment given on Day 2 to 9 of 2-week cycle.
  NOX66 dose of 800mg daily.
  Radiation treatment of 20Gy given over 5 daily fractions to selected target lesion/s for all cohorts.
  NOX66: NOX66 delivered as rectal suppository.
  Irradiation Therapy: Radiation per selected tumour lesion.
- Cohort 3 - NOX66 1200mg Daily: NOX66 administered on Days 1-16 and radiation treatment given on Day 2 to 9 of 2-week cycle.
  NOX66 dose of 1200mg daily.
  Radiation treatment of 20Gy given over 5 daily fractions to selected target lesion/s for all cohorts.
  NOX66: NOX66 delivered as rectal suppository.
  Irradiation Therapy: Radiation per selected tumour lesion.
- Cohort 4 - NOX66 1200mg Daily: NOX66 administered on Days 1-16 and radiation treatment given on Day 2 to 9 of 2-week cycle.
  NOX66 dose of 400mg daily.
  Radiation treatment of 20Gy given over 5 daily fractions to selected target lesion/s for all cohorts.
Period: Overall Study
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Started | 4 | 6 | 4 | 11
Completed | 4 | 3 | 4 | 5
Not Completed | 0 | 3 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Disease Progression | 0 | 0 | 0 | 3
Not completed — Death | 0 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 4 - NOX66 1200mg Daily: NOX66 administered on Days 1-16 and radiation treatment given on Day 2 to 9 of 2-week cycle.
  NOX66 dose of 1200mg daily.
  Radiation treatment of 20Gy given over 5 daily fractions to selected target lesion/s for all cohorts.
  NOX66: NOX66 delivered as rectal suppository.
  Irradiation Therapy: Radiation per selected tumour lesion.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily | Total
Number analyzed (Participants) | 4 | 6 | 4 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (8.06) | 68.5 (3.73) | 68.6 (5.25) | 70.6 (6.79) | 70.1 (6.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 4 | 6 | 4 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 6 | 4 | 11 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 0 | 0 | 1 | 0 | 0
  Georgia | 3 | 4 | 3 | 11 | 0
  Australia | 1 | 2 | 0 | 0 | 0
Diagnostic PSA level [Mean (Standard Deviation); unit: ng/mL] | 560.00 (579.828) | 222.38 (123.755) | 488.7 (0) | 154.0 (101.402) | 321.92 (258.950)
ECOG Performance Status at Screening [Count of Participants; unit: Participants]
  0 (Fully active) | 0 | 0 | 2 | 2 | 4
  1 (Ambulatory; No strenuous activity) | 4 | 6 | 2 | 9 | 21
  2 (Ambulatory; No work activity) | 0 | 0 | 0 | 0 | 0
  3 (Limited self-care) | 0 | 0 | 0 | 0 | 0
  4 (No self-care) | 0 | 0 | 0 | 0 | 0
  5 (Dead) | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events Including SAEs [Safety and Tolerability] of NOX66 Combined With Radiation Therapy at Multiple Timepoints
Description: Safety will be assessed through reported incidence of treatment emergent adverse events (AEs), including SAEs, dose limiting toxicities, AEs leading to withdrawal, events that are greater than CTCAE Version 4.03 Grade 2 in severity. Treatment emergent AEs are those with an onset on or after the initiation of therapy. Timepoints for AE /SAE assessment are Day 2 (start of radiation therapy treatment and one day after start of NOX66 treatment), Day 6, End of treatment (Day 16), Week 6, Week 12, and Week 24.
Time Frame: Day 2, Day 6, EOT (Day 16), Week 6, Week 12, and Week 24
Population: Safety population = all participants who received at least one dose of NOX66
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Participants
  Adverse events (AEs) | 4 | 5 | 2 | 9
  Treatment-emergent adverse events (TEAEs) | 4 | 5 | 2 | 9
  AEs that were DLTs | 0 | 0 | 0 | 0
  AEs leading to withdrawal | 0 | 0 | 0 | 0
  AEs that were greater than Grade 2 severity | 1 | 3 | 1 | 6
  Serious adverse events (SAEs) | 0 | 3 | 1 | 1

2. Primary Outcome: Assessment of Laboratory Results
Description: Mean change from Baseline in absolute value of safety laboratory results (haematology and biochemistry) assessed at End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
micromol/L
  Direct Bilirubin, Day 16 (micromol/L): number analyzed (Participants) | 3 | 4 | 3 | 11
  Direct Bilirubin, Day 16 (micromol/L) | 0.33 (0.583) | -0.78 (1.487) | -0.08 (0.415) | 0.16 (0.494)
  Direct Bilirubin, Week 6 (micromol/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Direct Bilirubin, Week 6 (micromol/L) | 0.33 (0.481) | -0.68 (0.864) | -0.26 (0.497) | -0.09 (0.320)
  Direct Bilirubin, Week 12 (micromol/L): number analyzed (Participants) | 4 | 3 | 3 | 11
  Direct Bilirubin, Week 12 (micromol/L) | -0.12 (0.872) | -0.46 (0.173) | -0.39 (0.521) | 0.19 (0.929)
  Direct Bilirubin, Week 24 (micromol/L): number analyzed (Participants) | 3 | 3 | 3 | 4
  Direct Bilirubin, Week 24 (micromol/L) | -0.03 (0.227) | -0.70 (0.735) | -0.26 (0.549) | 0.05 (0.135)
  Total Bilirubin, Day 16 (micromol/L) | 1.85 (2.229) | -0.35 (3.488) | -0.63 (2.447) | -0.26 (0.831)
  Total Bilirubin, Week 6 (micromol/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Total Bilirubin, Week 6 (micromol/L) | 2.45 (1.937) | 0.59 (0.897) | -0.48 (1.754) | -0.76 (1.120)
  Total Bilirubin, Week 12 (micromol/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Total Bilirubin, Week 12 (micromol/L) | -1.12 (3.749) | 0.90 (1.137) | 1.46 (2.034) | -0.92 (1.915)
  Total Bilirubin, Week 24 (micromol/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Total Bilirubin, Week 24 (micromol/L) | -1.35 (2.928) | -0.30 (0.567) | -1.43 (3.404) | -1.28 (2.483)
  Creatinine, Day 16 (micromol/L): number analyzed (Participants) | 4 | 6 | 3 | 11
  Creatinine, Day 16 (micromol/L) | 7.84 (38.883) | 4.64 (8.619) | 5.87 (8.122) | -2.90 (8.787)
  Creatinine, Week 6 (micromol/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Creatinine, Week 6 (micromol/L) | 15.77 (45.051) | -5.51 (9.603) | -2.33 (3.121) | 12.89 (21.919)
  Creatinine, Week 12 (micromol/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Creatinine, Week 12 (micromol/L) | -4.93 (11.097) | 16.32 (43.026) | -10.70 (0.300) | -10.63 (20.908)
  Creatinine, Week 24 (micromol/L): number analyzed (Participants) | 4 | 3 | 3 | 5
  Creatinine, Week 24 (micromol/L) | -5.98 (17.680) | -5.36 (9.032) | -8.90 (4.845) | -13.39 (16.696)

3. Primary Outcome: Assessment of ECG Results
Description: Mean change from Baseline in ECG intervals (msec) which are assessed at End of treatment (Day 16), Week 12, and Week 24.
Time Frame: Baseline to End of treatment (Day 16), Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
msec
  QT interval, Day 16: number analyzed (Participants) | 4 | 6 | 3 | 11
  QT interval, Day 16 | 24.1 (55.08) | -1.4 (33.29) | 9 (22.16) | 16.1 (33.53)
  QT interval, Week 12: number analyzed (Participants) | 4 | 4 | 3 | 11
  QT interval, Week 12 | 33.9 (68.59) | 4.8 (13.62) | -7 (23.67) | 7.6 (36.6)
  QT interval, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 5
  QT interval, Week 24 | 9.7 (34.76) | 4.8 (27.69) | 5.2 (25.62) | 9.2 (12.55)
  QTc interval, Day 16 | 19 (48.92) | 19.7 (32.1) | 11.1 (8.12) | 17.9 (40.32)
  QTc interval, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  QTc interval, Week 12 | 29.5 (30.88) | 17.0 (24.99) | 12.7 (6.39) | 15 (25.5)
  QTc interval, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 5
  QTc interval, Week 24 | 23.3 (29.57) | -2.6 (14.34) | 6.1 (11.55) | 0.8 (16.61)
  RR interval, Day 16: number analyzed (Participants) | 3 | 5 | 3 | 11
  RR interval, Day 16 | 23.4 (50.15) | -56.4 (123.08) | 7.6 (66.68) | 4.5 (212.55)
  RR interval, Week 12: number analyzed (Participants) | 3 | 3 | 3 | 11
  RR interval, Week 12 | 35.1 (201.4) | -11.6 (150.02) | -55.6 (140.05) | -20.1 (181.42)
  RR interval, Week 24: number analyzed (Participants) | 3 | 3 | 3 | 5
  RR interval, Week 24 | -54.4 (82.71) | 31.8 (59.97) | -17.2 (112.8) | 39.5 (38.78)

4. Primary Outcome: Assessment of Laboratory Results
Description: as for outcome 2
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: (g/L
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
(g/L
  Haemoglobin, Day 16 (g/L) | -0.5 (5.066) | -6.17 (9.579) | 1.5 (10.083) | -11.27 (8.956)
  Haemoglobin, Week 6 (g/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Haemoglobin, Week 6 (g/L) | -7.25 (13.598) | -8.50 (17.540) | -4.75 (10.532) | -11.27 (8.810)
  Haemoglobin, Week 12 (g/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Haemoglobin, Week 12 (g/L) | 11.00 (14.855) | 4.75 (21.140) | -6.00 (6.083) | -7.45 (15.247)
  Haemoglobin, Week 24 (g/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Haemoglobin, Week 24 (g/L) | 3.50 (6.608) | -2.00 (21.932) | -4.25 (6.397) | -14.60 (23.341)
  Mean Corpuscular Haemoglobin Concentration, Day 16 (g/L): number analyzed (Participants) | 4 | 5 | 3 | 11
  Mean Corpuscular Haemoglobin Concentration, Day 16 (g/L) | -16.75 (34.267) | -2.40 (8.989) | -4.33 (12.662) | 0.73 (3.062)
  Mean Corpuscular Haemoglobin Concentration, Week 6 (g/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Mean Corpuscular Haemoglobin Concentration, Week 6 (g/L) | 16.75 (38.922) | -4.25 (11.325) | 1.67 (2.082) | -2.00 (9.960)
  Mean Corpuscular Haemoglobin Concentration, Week 12 (g/L): number analyzed (Participants) | 4 | 3 | 3 | 11
  Mean Corpuscular Haemoglobin Concentration, Week 12 (g/L) | -13.00 (29.178) | -6.00 (8.888) | -1.33 (12.702) | -8.09 (28.339)
  Mean Corpuscular Haemoglobin Concentration, Week 24 (g/L): number analyzed (Participants) | 4 | 3 | 3 | 5
  Mean Corpuscular Haemoglobin Concentration, Week 24 (g/L) | -5.5 (31.754) | -2.67 (6.506) | -2.67 (8.622) | -0.80 (11.756)
  Albumin, Day 16 (g/L) | 0.80 (7.532) | -1.88 (5.518) | 0.34 (4.418) | -0.63 (4.785)
  Albumin, Week 6 (g/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Albumin, Week 6 (g/L) | -1.68 (2.538) | 4.58 (8.423) | -0.66 (7.579) | -3.88 (7.482)
  Albumin, Week 12 (g/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Albumin, Week 12 (g/L) | 0.10 (2.761) | 3.77 (8.070) | -1.01 (9.782) | -1.84 (5.678)
  Albumin, Week 24 (g/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Albumin, Week 24 (g/L) | -0.78 (3.497) | 3.77 (8.070) | -2.60 (8.497) | 0.58 (5.053)
  Total Protein, Day 16 (g/L) | 4.52 (6.700) | 0.36 (7.813) | -0.08 (7.023) | 0.23 (5.626)
  Total Protein, Week 6 (g/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Total Protein, Week 6 (g/L) | 4.04 (10.150) | 5.36 (7.813) | -0.08 (7.023) | -2.59 (9.247)
  Total Protein, Week 12 (g/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Total Protein, Week 12 (g/L) | 3.63 (5.397) | 7.44 (12.707) | 0.27 (15.883) | -0.68 (6.808)
  Total Protein, Week 24 (g/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Total Protein, Week 24 (g/L) | 1.43 (4.742) | 5.15 (14.853) | -2.68 (13.654) | 0.15 (6.919)

5. Primary Outcome: Assessment of Laboratory Results
Description: as for outcome 2
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: Percetange
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Percetange
  Haematocrit, Day 16 (%) | 2.13 (1.907) | -1.62 (3.029) | 0.80 (4.249) | -3.64 (3.281)
  Haematocrit, Week 6 (%): number analyzed (Participants) | 4 | 4 | 4 | 11
  Haematocrit, Week 6 (%) | 0.83 (1.489) | -2.23 (5.229) | -1.58 (3.040) | -3.25 (2.924)
  Haematocrit, Week 12 (%): number analyzed (Participants) | 4 | 4 | 3 | 11
  Haematocrit, Week 12 (%) | 6.83 (1.489) | -2.23 (5.229) | -1.58 (3.040) | -3.25 (2.924)
  Haematocrit, Week 24 (%): number analyzed (Participants) | 4 | 3 | 4 | 5
  Haematocrit, Week 24 (%) | 3.48 (5.067) | -0.40 (6.391) | -1.28 (2.313) | -4.42 (5.966)

6. Primary Outcome: Assessment of Laboratory Results
Description: as for outcome 2
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: 10^9cells/L
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
10^9cells/L
  Platelets, Day 16 (10^9/L) | -66.50 (50.849) | -37.00 (135.890) | -9.00 (121.351) | -45.45 (104.516)
  Platelets, Week 6 (10^9/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Platelets, Week 6 (10^9/L) | -81.50 (49.143) | -60.50 (86.002) | 83.00 (95.781) | -17.09 (58.066)
  Platelets, Week 12 (10^9/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Platelets, Week 12 (10^9/L) | -60.0 (101.278) | 36.25 (182.967) | -8.33 (129.894) | 28.36 (73.595)
  Platelets, Week 24 (10^9/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Platelets, Week 24 (10^9/L) | 86.75 (54.872) | -74.00 (65.818) | 34.75 (141.354) | 0.20 (79.998)
  White Blood Cells, Day 16 (10^9/L) | -2.99 (1.536) | 1.20 (1.694) | 2.10 (2.217) | -2.23 (2.269)
  White Blood Cells, Week 6 (10^9/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  White Blood Cells, Week 6 (10^9/L) | -3.13 (0.884) | -1.60 (1.632) | 3.42 (2.217) | -1.55 (1.543)
  White Blood Cells, Week 12 (10^9/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  White Blood Cells, Week 12 (10^9/L) | -2.93 (2.240) | 0.69 (2.565) | 4.62 (3.975) | -1.02 (2.331)
  White Blood Cells, Week 24 (10^9/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  White Blood Cells, Week 24 (10^9/L) | -2.42 (1.754) | -1.37 (1.086) | 2.63 (3.498) | -2.23 (2.676)
  Lymphocytes, Day 16 (10^9/L) | -0.57 (0.675) | -0.41 (0.770) | 0.35 (0.710) | -0.66 (1.113)
  Lymphocytes, Week 6 (10^9/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Lymphocytes, Week 6 (10^9/L) | 0.44 (0.497) | -0.75 (0.838) | 0.46 (0.901) | -0.39 (1.238)
  Lymphocytes, Week 12 (10^9/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Lymphocytes, Week 12 (10^9/L) | -0.38 (0.682) | -0.29 (0.792) | 0.24 (1.279) | -0.34 (1.175)
  Lymphocytes, Week 24 (10^9/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Lymphocytes, Week 24 (10^9/L) | -0.45 (0.768) | -1.25 (0.670) | 0.05 (0.854) | -0.71 (1.761)
  Neutrophils, Day 16 (10^9/L) | -0.02 (1.396) | 1.38 (1.926) | 1.47 (1.683) | -1.85 (1.926)
  Neutrophils, Week 6 (10^9/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Neutrophils, Week 6 (10^9/L) | -2.27 (0.641) | -0.77 (0.780) | 2.76 (1.050) | -1.50 (1.906)
  Neutrophils, Week 12 (10^9/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Neutrophils, Week 12 (10^9/L) | -2.00 (1.956) | 0.83 (1.466) | 4.27 (3.309) | -1.03 (2.245)
  Neutrophils, Week 24 (10^9/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Neutrophils, Week 24 (10^9/L) | -1.50 (0.776) | 0.11 (0.896) | 2.47 (2.607) | -2.33 (2.571)
  Monocytes, Day 16 (10^9/L) | -0.39 (0.623) | 0.19 (0.130) | 0.25 (0.200) | -0.06 (0.315)
  Monocytes, Week 6 (10^9/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Monocytes, Week 6 (10^9/L) | -0.42 (0622) | -0.13 (0.108) | 0.15 (0.137) | -0.05 (0.359)
  Monocytes, Week 12 (10^9/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Monocytes, Week 12 (10^9/L) | -0.55 (0.629) | 0.02 (0.310) | 0.12 (0.827) | 0.05 (0.396)
  Monocytes, Week 24 (10^9/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Monocytes, Week 24 (10^9/L) | -0.42 (0.565) | -0.11 (0.210) | 0.13 (0.541) | 0.29 (0.473)
  Eosinophils, Day 16 (10^9/L) | 0.00 (0.081) | 0.02 (0122) | 0.05 (0.097) | 0.05 (0.293)
  Eosinophils, Week 6 (10^9/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Eosinophils, Week 6 (10^9/L) | 0.01 (0.059) | 0.06 (0.120) | 0.04 (0.162) | -0.06 (0.176)
  Eosinophils, Week 12 (10^9/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Eosinophils, Week 12 (10^9/L) | 0.00 (0.081) | 0.04 (0.333) | -0.02 (0.076) | -0.07 (0.090)
  Eosinophils, Week 24 (10^9/L): number analyzed (Participants) | 4 | 3 | 3 | 5
  Eosinophils, Week 24 (10^9/L) | -0.02 (0.042) | -0.09 (0.148) | 0.00 (0.105) | -0.06 (0.119)
  Basophils, Day 16 (10^9/L): number analyzed (Participants) | 4 | 6 | 3 | 11
  Basophils, Day 16 (10^9/L) | -0.01 (0.010) | -0.01 (0.020) | 0.00 (0.006) | 0.00 (0.023)
  Basophils, Week 6 (10^9/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Basophils, Week 6 (10^9/L) | 0.30 (0.632) | -0.01 (0.010) | 0.02 (0.029) | 0.01 (0.019)
  Basophils, Week 12 (10^9/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Basophils, Week 12 (10^9/L) | 0.00 (0.005) | 0.03 (0.066) | 0.00 (0.006) | 0.00 (0.013)
  Basophils, Week 24 (10^9/L): number analyzed (Participants) | 4 | 3 | 3 | 5
  Basophils, Week 24 (10^9/L) | -0.01 (0.033) | -0.02 (0.006) | 0.00 (0.000) | -0.01 (0.020)

7. Primary Outcome: Assessment of Laboratory Results
Description: as for outcome 2
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: 10^12cells/L
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
10^12cells/L
  Red Blood Cells, Day 16 (10^12/L): number analyzed (Participants) | 4 | 6 | 3 | 4
  Red Blood Cells, Day 16 (10^12/L) | 0.05 (0.155) | -0.09 (0.526) | 0.25 (0.454) | -0.37 (0.445)
  Red Blood Cells, Week 6 (10^12/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Red Blood Cells, Week 6 (10^12/L) | -0.11 (0.415) | -0.34 (0.651) | -0.18 (0.599) | -0.32 (0.590)
  Red Blood Cells, Week 12 (10^12/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Red Blood Cells, Week 12 (10^12/L) | 0.55 (0.631) | 0.18 (0.7856) | -0.31 (0.176) | 0.01 (0.997)
  Red Blood Cells, Week 24 (10^12/L): number analyzed (Participants) | 4 | 3 | 3 | 5
  Red Blood Cells, Week 24 (10^12/L) | 0.09 (0.567) | -0.13 (0.766) | -0.28 (0.350) | -0.32 (0.887)

8. Primary Outcome: Assessment of Laboratory Results
Description: as for outcome 2
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
U/L
  ALP, Day 16 (U/L) | 57.53 (83.556) | -35.34 (142460) | -11.53 (13.814) | -33.68 (176.815)
  ALP, Week 6 (U/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  ALP, Week 6 (U/L) | 228.28 (230.132) | -95.55 (193.289) | 3.60 (31.794) | -11.73 (184.158)
  ALP, Week 12 (U/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  ALP, Week 12 (U/L) | 261.98 (220.518) | -142.00 (225.295) | -17.00 (7.791) | 144.01 (250.644)
  ALP, Week 24 (U/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  ALP, Week 24 (U/L) | 271.30 (172.254) | -167.33 (328.804) | -16.10 (12.928) | -26.66 (27.916)
  ALT, Day 16 (U/L) | 0.56 (2.380) | 0.02 (13.231) | 0.13 (2.347) | -0.65 (8.070)
  ALT, Week 6 (U/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  ALT, Week 6 (U/L) | 0.93 (3.621) | -1.24 (4.199) | -0.28 (6.779) | 0.00 (8.286)
  ALT, Week 12 (U/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  ALT, Week 12 (U/L) | 0.40 (2.637) | -5.93 (15.796) | -1.80 (6.948) | -4.58 (11.113)
  ALT, Week 24 (U/L): number analyzed (Participants) | 4 | 3 | 4 | 11
  ALT, Week 24 (U/L) | -0.96 (1.077) | 0.56 (4.801) | -0.85 (2.420) | -1.11 (2.961)
  AST, Day 16 (U/L): number analyzed (Participants) | 4 | 6 | 4 | 5
  AST, Day 16 (U/L) | 2.14 (0.869) | 5.87 (6.867) | 0.00 (0.000) | -4.59 (9.102)
  AST, Week 6 (U/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  AST, Week 6 (U/L) | 5.24 (6.508) | 0.74 (2.413) | 1.08 (2.045) | -4.87 (6.70)
  AST, Week 12 (U/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  AST, Week 12 (U/L) | 2.14 (1.919) | -1.26 (5.592) | 4.03 (1.861) | 5.03 (23.916)
  AST, Week 24 (U/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  AST, Week 24 (U/L) | 6.64 (6.137) | -3.42 (8.199) | -0.78 (2.382) | -2.08 (3.281)

9. Primary Outcome: Assessment of Laboratory Results
Description: as for outcome 2
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
fL
  Mean Corpuscular Volume, Day 16 (fL) | 4.10 (6.968) | -1.58 (5.278) | -2.55 (6.125) | -0.26 (4.713)
  Mean Corpuscular Volume, Week 6 (fL): number analyzed (Participants) | 4 | 4 | 4 | 11
  Mean Corpuscular Volume, Week 6 (fL) | 4.60 (7.124) | 2.40 (3.713) | -0.53 (73.486) | 0.45 (7.486)
  Mean Corpuscular Volume, Week 12 (fL): number analyzed (Participants) | 4 | 4 | 3 | 11
  Mean Corpuscular Volume, Week 12 (fL) | 3.50 (3.696) | 1.10 (3.451) | 2.53 (4.957) | -1.05 (5.025)
  Mean Corpuscular Volume, Week 24 (fL): number analyzed (Participants) | 4 | 3 | 4 | 5
  Mean Corpuscular Volume, Week 24 (fL) | 5.05 (6.357) | 2.03 (1.704) | 1.30 (4.577) | -2.26 (8.719)

10. Primary Outcome: Assessment of Laboratory Results
Description: as for outcome 2
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
pg
  Mean Corpuscular Haemoglobin, Day 16 (pg) | 0.13 (0.862) | -0.97 (1.632) | -1.15 (1.353) | 0.22 (2.586)
  Mean Corpuscular Haemoglobin, Week 6 (pg): number analyzed (Participants) | 4 | 4 | 4 | 11
  Mean Corpuscular Haemoglobin, Week 6 (pg) | 0.23 (0.862) | 0.33 (1.109) | 0.05 (2.603) | -0.17 (1.797)
  Mean Corpuscular Haemoglobin, Week 12 (pg): number analyzed (Participants) | 4 | 4 | 3 | 11
  Mean Corpuscular Haemoglobin, Week 12 (pg) | 0.23 (1.056) | 0.05 (1.015) | 0.83 (2.403) | -2.05 (4.155)
  Mean Corpuscular Haemoglobin, Week 24 (pg): number analyzed (Participants) | 4 | 3 | 4 | 5
  Mean Corpuscular Haemoglobin, Week 24 (pg) | 1.35 (1.212) | 0.40 (0.985) | 1.33 (3.822) | -0.76 (3.062)

11. Secondary Outcome: Change of Target Lesions in Participants According to RECIST 1.1 Criteria
Description: RECIST response in target irradiated and non-irradiated lesions based on radiographic CT/MRI scan. RECIST 1.1 criteria are Complete Response (CR), Partial Response (PR), Stable Disease(SD) and Progressive Disease (PD). Not Applicable (NA) indicates that a participant did not have measurable target lesions at Screening.
Time Frame: Week 6, Week 12, and Week 24
Population: Efficacy population = all patients who completed radiation therapy with at least seven days of NOX66 treatment
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3 NOX66 1200mg Daily; Cohort 4 - NOX66 1200mg Daily: NOX66 administered on Days 1-16 and radiation treatment given on Day 2 to 9 of 2-week cycle.
  NOX66 dose of 1200mg daily.
  Radiation treatment of 20Gy given over 5 daily fractions to selected target lesion/s for all cohorts.
  NOX66: NOX66 delivered as rectal suppository.
  Irradiation Therapy: Radiation per selected tumour lesion.
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Participants
  Week 6: Complete Response (CR) | 0 | 0 | 0 | 0
  Week 6: Partial Response (PR) | 0 | 0 | 0 | 1
  Week 6: Stable Disease (SD) | 4 | 4 | 4 | 8
  Week 6: Progressive Disease (PD) | 0 | 0 | 0 | 0
  Week 6: Not Evaluable (NE) | 0 | 2 | 0 | 0
  Week 6: Not Applicable (NA) | 0 | 0 | 0 | 2
  Week 12: Complete Response (CR) | 0 | 0 | 0 | 0
  Week 12: Partial Response (PR) | 0 | 1 | 0 | 2
  Week 12: Stable Disease (SD) | 4 | 2 | 3 | 5
  Week 12: Progressive Disease (PD) | 0 | 1 | 0 | 0
  Week 12: Not Evaluable (NE) | 0 | 2 | 1 | 2
  Week 12: Not Applicable (NA) | 0 | 0 | 0 | 2
  Week 24: Complete Response (CR) | 0 | 0 | 0 | 0
  Week 24: Partial Response (PR) | 0 | 1 | 0 | 1
  Week 24: Stable Disease (SD) | 3 | 2 | 3 | 2
  Week 24: Progressive Disease (PD) | 0 | 0 | 0 | 0
  Week 24: Not Evaluable (NE) | 1 | 3 | 1 | 6
  Week 24: Not Applicable (NA) | 0 | 0 | 0 | 2

12. Secondary Outcome: Change of Non-Target Lesions in Participants According to RECIST 1.1 Criteria
Description: RECIST 1.1 assessment of response in Non-Target Lesions as Complete Response (CR), Non-CR/Non-PD, or Progressive Disease (PD). Not Applicable (NA) signifies that the participant did not have non-target lesions at Screening.
Time Frame: Week 6, Week 12, and Week 24
Population: Efficacy population = all patients who completed radiation therapy with at least seven days of NOX66 treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Participants
  Week 6: Complete Response (CR) | 0 | 0 | 0 | 0
  Week 6: Non-CR/Non-PD | 4 | 5 | 3 | 7
  Week 6: Progressive Disease (PD) | 0 | 0 | 0 | 0
  Week 6: Not Evaluable (NE) | 0 | 0 | 0 | 4
  Week 6: Not Applicable (NA) | 0 | 1 | 1 | 0
  Week 12: Complete Response (CR) | 0 | 0 | 1 | 0
  Week 12: Non-CR/Non-PD | 4 | 4 | 2 | 7
  Week 12: Progressive Disease (PD) | 0 | 1 | 0 | 0
  Week 12: Not Evaluable (NE) | 0 | 0 | 0 | 4
  Week 12: Not Applicable (NA) | 0 | 1 | 1 | 0
  Week 24: Complete Response (CR) | 1 | 0 | 1 | 1
  Week 24: Non-CR/Non-PD | 2 | 4 | 2 | 6
  Week 24: Progressive Disease (PD) | 1 | 1 | 0 | 1
  Week 24: Not Evaluable (NE) | 0 | 0 | 0 | 3
  Week 24: Not Applicable (NA) | 0 | 1 | 1 | 0

13. Secondary Outcome: Overall Response According to RECIST 1.1 Criteria
Description: Overall RECIST 1.1 response based on combined assessment criteria for target, non-target and new lesions as Complete Response (CR), Partial Response (PR), Stable Disease(SD), or Progressive Disease (PD)
Time Frame: From enrolment up to Week 6, Week 12, and Week 24
Population: Efficacy population = all patients who completed radiation therapy with at least seven days of NOX66 treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Participants
  Week 6: Complete Response (CR) | 0 | 0 | 0 | 0
  Week 6: Partial Response (PR) | 0 | 0 | 0 | 1
  Week 6: Stable Disease (SD) | 4 | 3 | 4 | 9
  Week 6: Progressive Disease (PD) | 0 | 1 | 0 | 0
  Week 6: Not Evaluable (NE) | 0 | 2 | 0 | 1
  Week 12: Complete Response (CR) | 0 | 0 | 0 | 0
  Week 12: Partial Response (PR) | 0 | 1 | 0 | 2
  Week 12: Stable Disease (SD) | 3 | 2 | 3 | 6
  Week 12: Progressive Disease (PD) | 1 | 1 | 0 | 0
  Week 12: Not Evaluable (NE) | 0 | 2 | 1 | 3
  Week 24: Complete Response (CR) | 0 | 0 | 0 | 0
  Week 24: Partial Response (PR) | 0 | 1 | 0 | 0
  Week 24: Stable Disease (SD) | 2 | 2 | 3 | 2
  Week 24: Progressive Disease (PD) | 1 | 0 | 0 | 3
  Week 24: Not Evaluable (NE) | 1 | 3 | 1 | 6

14. Secondary Outcome: Change in Overall Pain Score Using the Brief Pain Inventory - Short Form (BPI-SF)
Description: Percentage change from baseline in overall pain score based on responses to the BPI-SF, which is scored from 0 to 10, with 0 = no pain and 10 = the most severe pain imaginable.
Time Frame: From enrolment up to Day 16, Week 6, Week 12, and Week 24
Population: Efficacy population = all patients who completed radiation therapy with at least seven days of NOX66 treatment
Measure: Mean (Standard Deviation); unit: Percentage change from baseline in score
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Percentage change from baseline in score
  Day 16: number analyzed (Participants) | 4 | 6 | 4 | 10
  Day 16 | -52.186 (56.6238) | 32.737 (103.7459) | 3.6 (32.30) | -37.2 (37.92)
  Week 6: number analyzed (Participants) | 4 | 4 | 4 | 10
  Week 6 | -58.954 (40.1178) | -47.815 (35.0069) | -44.1 (44.36) | -41.8 (42.28)
  Week 12: number analyzed (Participants) | 4 | 4 | 3 | 10
  Week 12 | -55.830 (52.9611) | -29.175 (82.3088) | 42.8 (44.46) | -37.0 (47.51)
  Week 24: number analyzed (Participants) | 4 | 3 | 4 | 5
  Week 24 | 10.786 (46.4994) | -80.992 (32.9233) | -38.4 (35.16) | -68.6 (49.04)

15. Secondary Outcome: Change in Prostate Specific Antigen (PSA) Levels
Description: Percentage change from baseline in serum PSA levels (ng/mL) at Week 6, Week 12, and Week 24
Time Frame: From enrolment up to Week 6, Week 12, and Week 24
Population: Efficacy population = all patients who completed radiation therapy with at least seven days of NOX66 treatment
Measure: Mean (Standard Deviation); unit: Percentage change from baseline in PSA
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Percentage change from baseline in PSA
  Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Week 6 | 17.79 (42.116) | -46.67 (27.358) | 0.29 (41.424) | -19.49 (52.989)
  Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Week 12 | 35.75 (31.610) | -53.26 (31.766) | 14.82 (138.637) | -310 (73.373)
  Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Week 24 | 333.51 (357.538) | -14.85 (62.764) | 374.20 (518.309) | 64.86 (195.334)

16. Secondary Outcome: Change of ECOG Performance Status
Description: Assessment of patient via ECOG Performance Status, which has a scale scored from 0 (Fully Active) to 5 (Dead).
Time Frame: From enrolment up to Week 6, Week 12, and Week 24
Population: Efficacy population = all patients who completed radiation therapy with at least seven days of NOX66 treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Participants
  Screening: 0 (Fully active) | 0 | 0 | 2 | 2
  Screening: 1 (Ambulatory; No strenuous activity) | 4 | 6 | 2 | 9
  Screening: 2 (Ambulatory; No work activity) | 0 | 0 | 0 | 0
  Screening: 3 (Limited self-care) | 0 | 0 | 0 | 0
  Screening: 4 (No self-care) | 0 | 0 | 0 | 0
  Screening: 5 (Dead) | 0 | 0 | 0 | 0
  Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Week 6: 0 (Fully active) | 0 | 1 | 2 | 1
  Week 6: 1 (Ambulatory; No strenuous activity) | 4 | 3 | 1 | 7
  Week 6: 2 (Ambulatory; No work activity) | 0 | 0 | 1 | 3
  Week 6: 3 (Limited self-care) | 0 | 0 | 0 | 0
  Week 6: 4 (No self-care) | 0 | 0 | 0 | 0
  Week 6: 5 (Dead) | 0 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 4 | 4 | 3 | 11
  Week 12: 0 (Fully active) | 0 | 2 | 2 | 2
  Week 12: 1 (Ambulatory; No strenuous activity) | 4 | 1 | 1 | 5
  Week 12: 2 (Ambulatory; No work activity) | 0 | 1 | 0 | 2
  Week 12: 3 (Limited self-care) | 0 | 0 | 0 | 1
  Week 12: 4 (No self-care) | 0 | 0 | 0 | 1
  Week 12: 5 (Dead) | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 4 | 4 | 4 | 5
  Week 24: 0 (Fully active) | 0 | 2 | 2 | 2
  Week 24: 1 (Ambulatory; No strenuous activity) | 3 | 1 | 1 | 1
  Week 24: 2 (Ambulatory; No work activity) | 1 | 0 | 0 | 1
  Week 24: 3 (Limited self-care) | 0 | 0 | 1 | 1
  Week 24: 4 (No self-care) | 0 | 0 | 0 | 0
  Week 24: 5 (Dead) | 0 | 1 | 0 | 0

17. Secondary Outcome: Assessment of Change in Physical Appearance (Physical Exam) by Measuring HEENT, Gastrointestinal, Abdominal Status at Multiple Timepoints
Description: Assessment of patient via physical exam comparing Day 2, End of Treatment (Day 16), Week 6, Week 12, and Week 24 to baseline. Physical exam included abdominal, cardiovascular, dermatologic, gastrointestinal, genitourinary, HEENT (head, eyes, ears, nose, throat), lymphatic, musculoskeletal, neurological, other, and pulmonary exams.
Time Frame: From enrolment up to Day 2, End of Treatment (Day 16), Week 6, Week 12, and Week 24
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
Participants
  Abdominal Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  Abdominal Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Abdominal Exam, Day 2: No change | 4 | 5 | 4 | 11
  Abdominal Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  Abdominal Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Abdominal Exam, Day 16: No change | 4 | 6 | 4 | 11
  Abdominal Exam, Day 16: Worsened | 0 | 0 | 0 | 0
  Abdominal Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Abdominal Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Abdominal Exam, Week 6: No change | 4 | 4 | 4 | 11
  Abdominal Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Abdominal Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Abdominal Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Abdominal Exam, Week 12: No change | 4 | 4 | 4 | 11
  Abdominal Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Abdominal Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Abdominal Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Abdominal Exam, Week 24: No change | 4 | 3 | 4 | 11
  Abdominal Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  Cardiovascular Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  Cardiovascular Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Cardiovascular Exam, Day 2: No change | 4 | 5 | 4 | 11
  Cardiovascular Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  Cardiovascular Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Cardiovascular Exam, Day 16: No change | 4 | 6 | 4 | 11
  Cardiovascular Exam, Day 16: Worsened | 0 | 0 | 0 | 0
  Cardiovascular Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Cardiovascular Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Cardiovascular Exam, Week 6: No change | 4 | 4 | 4 | 11
  Cardiovascular Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Cardiovascular Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Cardiovascular Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Cardiovascular Exam, Week 12: No change | 4 | 4 | 4 | 11
  Cardiovascular Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Cardiovascular Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Cardiovascular Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Cardiovascular Exam, Week 24: No change | 4 | 3 | 4 | 11
  Cardiovascular Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  Dermatologic Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  Dermatologic Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Dermatologic Exam, Day 2: No change | 4 | 5 | 4 | 11
  Dermatologic Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  Dermatologic Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Dermatologic Exam, Day 16: No change | 4 | 5 | 4 | 11
  Dermatologic Exam, Day 16: Worsened | 0 | 1 | 0 | 0
  Dermatologic Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Dermatologic Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Dermatologic Exam, Week 6: No change | 4 | 4 | 4 | 11
  Dermatologic Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Dermatologic Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Dermatologic Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Dermatologic Exam, Week 12: No change | 4 | 4 | 4 | 11
  Dermatologic Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Dermatologic Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Dermatologic Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Dermatologic Exam, Week 24: No change | 4 | 3 | 4 | 11
  Dermatologic Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  Gastrointestinal Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  Gastrointestinal Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Gastrointestinal Exam, Day 2: No change | 4 | 4 | 4 | 11
  Gastrointestinal Exam, Day 2: Worsened | 0 | 1 | 0 | 0
  Gastrointestinal Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Gastrointestinal Exam, Day 16: No change | 4 | 5 | 4 | 11
  Gastrointestinal Exam, Day 16: Worsened | 0 | 1 | 0 | 0
  Gastrointestinal Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Gastrointestinal Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Gastrointestinal Exam, Week 6: No change | 4 | 4 | 4 | 11
  Gastrointestinal Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Gastrointestinal Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Gastrointestinal Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Gastrointestinal Exam, Week 12: No change | 4 | 4 | 4 | 11
  Gastrointestinal Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Gastrointestinal Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Gastrointestinal Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Gastrointestinal Exam, Week 24: No change | 4 | 3 | 4 | 11
  Gastrointestinal Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  Genitourinary Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  Genitourinary Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Genitourinary Exam, Day 2: No change | 4 | 5 | 4 | 11
  Genitourinary Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  Genitourinary Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Genitourinary Exam, Day 16: No change | 4 | 5 | 4 | 11
  Genitourinary Exam, Day 16: Worsened | 0 | 1 | 0 | 0
  Genitourinary Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Genitourinary Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Genitourinary Exam, Week 6: No change | 4 | 4 | 4 | 11
  Genitourinary Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Genitourinary Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Genitourinary Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Genitourinary Exam, Week 12: No change | 4 | 4 | 4 | 11
  Genitourinary Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Genitourinary Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Genitourinary Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Genitourinary Exam, Week 24: No change | 4 | 3 | 4 | 11
  Genitourinary Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  HEENT Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  HEENT Exam, Day 2: Improved | 0 | 0 | 0 | 0
  HEENT Exam, Day 2: No change | 4 | 5 | 4 | 11
  HEENT Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  HEENT Exam, Day 16: Improved | 0 | 0 | 0 | 0
  HEENT Exam, Day 16: No change | 4 | 6 | 4 | 11
  HEENT Exam, Day 16: Worsened | 0 | 0 | 0 | 0
  HEENT Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  HEENT Exam, Week 6: Improved | 0 | 0 | 0 | 0
  HEENT Exam, Week 6: No change | 4 | 4 | 4 | 11
  HEENT Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  HEENT Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  HEENT Exam, Week 12: Improved | 0 | 0 | 0 | 0
  HEENT Exam, Week 12: No change | 4 | 4 | 4 | 11
  HEENT Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  HEENT Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  HEENT Exam, Week 24: Improved | 0 | 0 | 0 | 0
  HEENT Exam, Week 24: No change | 4 | 3 | 4 | 11
  HEENT Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  Lymphatic Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  Lymphatic Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Lymphatic Exam, Day 2: No change | 4 | 5 | 4 | 11
  Lymphatic Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  Lymphatic Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Lymphatic Exam, Day 16: No change | 4 | 6 | 4 | 11
  Lymphatic Exam, Day 16: Worsened | 0 | 0 | 0 | 0
  Lymphatic Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Lymphatic Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Lymphatic Exam, Week 6: No change | 4 | 4 | 4 | 11
  Lymphatic Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Lymphatic Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Lymphatic Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Lymphatic Exam, Week 12: No change | 4 | 4 | 4 | 11
  Lymphatic Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Lymphatic Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Lymphatic Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Lymphatic Exam, Week 24: No change | 4 | 3 | 4 | 11
  Lymphatic Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  Musculoskeletal Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  Musculoskeletal Exam, Day 2: Improved | 0 | 1 | 0 | 0
  Musculoskeletal Exam, Day 2: No change | 4 | 4 | 3 | 11
  Musculoskeletal Exam, Day 2: Worsened | 0 | 0 | 1 | 0
  Musculoskeletal Exam, Day 16: Improved | 0 | 1 | 0 | 0
  Musculoskeletal Exam, Day 16: No change | 4 | 5 | 3 | 11
  Musculoskeletal Exam, Day 16: Worsened | 0 | 0 | 1 | 0
  Musculoskeletal Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Musculoskeletal Exam, Week 12: Improved | 0 | 0 | 0 | 1
  Musculoskeletal Exam, Week 12: No change | 4 | 3 | 3 | 10
  Musculoskeletal Exam, Week 12: Worsened | 0 | 1 | 1 | 0
  Musculoskeletal Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Musculoskeletal Exam, Week 6: Improved | 0 | 1 | 0 | 0
  Musculoskeletal Exam, Week 6: No change | 4 | 3 | 3 | 11
  Musculoskeletal Exam, Week 6: Worsened | 0 | 0 | 1 | 0
  Musculoskeletal Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Musculoskeletal Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Musculoskeletal Exam, Week 24: No change | 4 | 3 | 3 | 11
  Musculoskeletal Exam, Week 24: Worsened | 0 | 0 | 1 | 0
  Neurological Exam, Day 2: number analyzed (Participants) | 3 | 5 | 4 | 11
  Neurological Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Neurological Exam, Day 2: No change | 3 | 5 | 4 | 11
  Neurological Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  Neurological Exam, Day 16: number analyzed (Participants) | 3 | 6 | 4 | 11
  Neurological Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Neurological Exam, Day 16: No change | 3 | 6 | 4 | 11
  Neurological Exam, Day 16: Worsened | 0 | 0 | 0 | 0
  Neurological Exam, Week 6: number analyzed (Participants) | 3 | 4 | 4 | 11
  Neurological Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Neurological Exam, Week 6: No change | 3 | 4 | 4 | 11
  Neurological Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Neurological Exam, Week 12: number analyzed (Participants) | 3 | 4 | 4 | 11
  Neurological Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Neurological Exam, Week 12: No change | 3 | 4 | 4 | 11
  Neurological Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Neurological Exam, Week 24: number analyzed (Participants) | 3 | 3 | 4 | 11
  Neurological Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Neurological Exam, Week 24: No change | 3 | 3 | 4 | 11
  Neurological Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  Other Exam, Day 2: number analyzed (Participants) | 1 | 3 | 1 | 6
  Other Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Other Exam, Day 2: No change | 1 | 3 | 1 | 6
  Other Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  Other Exam, Day 16: number analyzed (Participants) | 1 | 3 | 1 | 6
  Other Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Other Exam, Day 16: No change | 1 | 3 | 1 | 6
  Other Exam, Day 16: Worsened | 0 | 0 | 0 | 0
  Other Exam, Week 6: number analyzed (Participants) | 1 | 2 | 1 | 6
  Other Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Other Exam, Week 6: No change | 1 | 2 | 1 | 6
  Other Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Other Exam, Week 12: number analyzed (Participants) | 1 | 2 | 1 | 6
  Other Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Other Exam, Week 12: No change | 1 | 2 | 1 | 6
  Other Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Other Exam, Week 24: number analyzed (Participants) | 1 | 2 | 1 | 6
  Other Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Other Exam, Week 24: No change | 1 | 2 | 1 | 6
  Other Exam, Week 24: Worsened | 0 | 0 | 0 | 0
  Pulmonary Exam, Day 2: number analyzed (Participants) | 4 | 5 | 4 | 11
  Pulmonary Exam, Day 2: Improved | 0 | 0 | 0 | 0
  Pulmonary Exam, Day 2: No change | 4 | 5 | 4 | 11
  Pulmonary Exam, Day 2: Worsened | 0 | 0 | 0 | 0
  Pulmonary Exam, Day 16: Improved | 0 | 0 | 0 | 0
  Pulmonary Exam, Day 16: No change | 4 | 6 | 4 | 11
  Pulmonary Exam, Day 16: Worsened | 0 | 0 | 0 | 0
  Pulmonary Exam, Week 6: number analyzed (Participants) | 4 | 4 | 4 | 11
  Pulmonary Exam, Week 6: Improved | 0 | 0 | 0 | 0
  Pulmonary Exam, Week 6: No change | 4 | 4 | 4 | 11
  Pulmonary Exam, Week 6: Worsened | 0 | 0 | 0 | 0
  Pulmonary Exam, Week 12: number analyzed (Participants) | 4 | 4 | 4 | 11
  Pulmonary Exam, Week 12: Improved | 0 | 0 | 0 | 0
  Pulmonary Exam, Week 12: No change | 4 | 4 | 4 | 11
  Pulmonary Exam, Week 12: Worsened | 0 | 0 | 0 | 0
  Pulmonary Exam, Week 24: number analyzed (Participants) | 4 | 3 | 4 | 11
  Pulmonary Exam, Week 24: Improved | 0 | 0 | 0 | 0
  Pulmonary Exam, Week 24: No change | 4 | 3 | 4 | 11
  Pulmonary Exam, Week 24: Worsened | 0 | 0 | 0 | 0

18. Primary Outcome: Assessment of Laboratory Results
Description: as for outcome 2
Time Frame: From Baseline to End of Treatment (Day 16), Week 6, Week 12, and Week 24.
Population: Safety population = all patients who received at least one dose of NOX66
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
Number analyzed (Participants) | 4 | 6 | 4 | 11
mmol/L
  Sodium, Day 16 (mmol/L) | -2.10 (3.075) | -0.65 (2.620) | -0.180 (2.917) | -1.52 (3.257)
  Sodium, Week 6 (mmol/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Sodium, Week 6 (mmol/L) | -2.60 (5.411) | 1.25 (3.573) | 0.93 (3.645) | -2.09 (3.198)
  Sodium, Week 12 (mmol/L): number analyzed (Participants) | 4 | 4 | 3 | 11
  Sodium, Week 12 (mmol/L) | -1.83 (4.664) | 1.83 (1.756) | 1.07 (2.901) | -1.43 (4.052)
  Sodium, Week 24 (mmol/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Sodium, Week 24 (mmol/L) | -2.73 (1.977) | 2.23 (4.450) | 1.45 (3.779) | 0.60 (1.056)
  Potassium, Day 16 (mmol/L) | -0.38 (0.078) | -0.27 (0.222) | -0.25 (0.311) | 0.03 (0.676)
  Potassium, Week 6 (mmol/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Potassium, Week 6 (mmol/L) | -0.39 (0.401) | -0.32 (0.495) | -0.19 (0.694) | -0.14 (0.736)
  Potassium, Week 12 (mmol/L): number analyzed (Participants) | 4 | 4 | 4 | 11
  Potassium, Week 12 (mmol/L) | -0.19 (0.388) | -0.12 (0.662) | 0.24 (0.392) | -0.09 (0.710)
  Potassium, Week 24 (mmol/L): number analyzed (Participants) | 4 | 3 | 4 | 5
  Potassium, Week 24 (mmol/L) | -0.23 (0.301) | -0.01 (0.609) | 0.10 (0.612) | 0.35 (0.689)
  Calcium, Day 16 (mmol/L): number analyzed (Participants) | 4 | 6 | 3 | 10
  Calcium, Day 16 (mmol/L) | -0.05 (0.058) | -0.20 (0.201) | -0.07 (0.101) | -0.08 (0.507)
  Calcium, Week 6 (mmol/L): number analyzed (Participants) | 4 | 4 | 3 | 10
  Calcium, Week 6 (mmol/L) | -0.31 (0.403) | 0.01 (0.340) | -0.15 (0.159) | -0.06 (0.504)
  Calcium, Week 12 (mmol/L): number analyzed (Participants) | 4 | 4 | 3 | 10
  Calcium, Week 12 (mmol/L) | 0.03 (0.144) | -0.39 (0.460) | -0.09 (0.075) | -0.19 (0.451)
  Calcium, Week 24 (mmol/L): number analyzed (Participants) | 4 | 3 | 3 | 4
  Calcium, Week 24 (mmol/L) | 0.36 (0.415) | -0.06 (0.191) | 0.00 (0.084) | -0.07 (0.574)

ADVERSE EVENTS:
Time Frame: Individual subjects = 9 months. Entire study = 19 months.
Arm/Group | Cohort 1 - NOX66 400mg Daily | Cohort 2 - NOX66 800mg Daily | Cohort 3 - NOX66 1200mg Daily | Cohort 4 - NOX66 1200mg Daily
All-Cause Mortality (participants affected / at risk) | 0/4 | 3/6 | 0/4 | 1/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 3/6 | 1/4 | 1/11
Other Adverse Events (participants affected / at risk) | 4/4 | 5/6 | 2/4 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - NOX66 400mg Daily (N=4) | Cohort 2 - NOX66 800mg Daily (N=6) | Cohort 3 - NOX66 1200mg Daily (N=4) | Cohort 4 - NOX66 1200mg Daily (N=11)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - NOX66 400mg Daily (N=4) | Cohort 2 - NOX66 800mg Daily (N=6) | Cohort 3 - NOX66 1200mg Daily (N=4) | Cohort 4 - NOX66 1200mg Daily (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0) | 7 (12)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (2) | 6 (12)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 120 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT03307629/Prot_SAP_000.pdf